CLINICAL TRIAL: NCT04305327
Title: A Phase 3, Randomised, Double-blind, Multi-centre Trial to Evaluate the Efficacy, Safety, and Tolerability of Brodalumab Treatment Compared to Placebo and Ustekinumab in Adolescent Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: Efficacy and Safety of Brodalumab in Adolescents From 12 to 17 Years of Age With Moderate-to-severe Plaque Psoriasis
Acronym: EMBRACE 1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Early terminated due to difficulty recruiting participants
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0160-1396; 2019-001868-30 (EudraCT Number); U1111-1282-4459 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind until Week 12, where the primary endpoint is assessed. Open-label active comparator treatment from Week 0 to Week 52, but with blinded outcomes assessor throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Brodalumab (Experimental): Brodalumab for 52 weeks. The dose will be determined by the participant's body weight.
  Interventions: Drug: Brodalumab
- Ustekinumab (Active Comparator): Ustekinumab for 52 weeks. The dose will be determined by the participant's body weight.
  Interventions: Drug: Ustekinumab
- Placebo/brodalumab (Placebo Comparator): Placebo for the first 12 weeks and brodalumab for the following 40 weeks. The dose will be determined by the participant's body weight.
  Interventions: Drug: Brodalumab; Drug: Placebo
- Placebo/ustekinumab (Placebo Comparator): Placebo for the first 12 weeks and ustekinumab for the following 40 weeks. The dose will be determined by the participant's body weight.
  Interventions: Drug: Ustekinumab; Drug: Placebo

INTERVENTIONS:
Drug: Brodalumab — Solution for subcutaneous injection.
  Other Names: Kyntheum®
  Arms: Brodalumab; Placebo/brodalumab
Drug: Ustekinumab — Solution for subcutaneous injection.
  Other Names: Stelara®
  Arms: Placebo/ustekinumab; Ustekinumab
Drug: Placebo — The placebo solution is similar to the active brodalumab solution except that it does not contain any active substance.
  Arms: Placebo/brodalumab; Placebo/ustekinumab

SUMMARY:
The study will investigate the efficacy and safety compared to placebo and the safety compared to ustekinumab of brodalumab in adolescents with moderate to severe plaque psoriasis. The study will also investigate if brodalumab affects development of vaccination-induced immune responses.

The study will run over 62-64 weeks (including screening, treatment, and safety follow-up) for each participant, but with the primary endpoint measured at Week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject was diagnosed with chronic plaque psoriasis at least 6 months before randomisation.
* Subject has a diagnosis of moderate-to-severe plaque psoriasis as defined by PASI ≥12, sPGA ≥3, and body surface area ≥10% at screening and at baseline.
* Subject, in whom topical therapy is not adequate, and who is a candidate for systemic therapy.
* Subject has no evidence of active or latent tuberculosis according to local standard of care.

Key Exclusion Criteria:

* Subject is diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions (e.g., eczema).
* Subject has been vaccinated with a tetanus toxoid-containing vaccine ≤18 months prior to first dose of investigational medicinal product (IMP). For EU and UK: Subject has been vaccinated with a TT-containing vaccine within 5 years prior to the first dose of IMP.
* Subject has developed or experienced either Guillian-Barre syndrome, encephalopathy, Arthus-type hypersensitivity, or severe allergic reactions in connection with previous Tdap or Td vaccine.
* Subject with chronic or recurrent infections, or active infection, systemically treated within 4 weeks prior to first dose of IMP.
* Subject has a known history of Crohn's disease.
* Subject has any active malignancy or a history of any malignancy within 5 years.
* Subject has a history of suicidal behaviour and has suicidal ideation with some intent to act or specific plan and intent.
* Subject has a history of depressive disorder with severe episode(s) within the last 2 years.
* Subject has received anti-IL-12/23p40 for less than 12 months prior to the first dose of IMP or has previously no response to anti-IL-12/23p40 therapy.
* Subject has previously received anti-IL-17 therapy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (31):
- Belgium (2):
  - LEO Pharma Investigational Site, Brussels
  - LEO Pharma Investigational Site, Liège
- LEO Pharma Investigational Site, Toulouse, France
- Germany (8):
  - LEO Pharma Investigational Site, Bad Bentheim
  - LEO Pharma Investigational Site, Essen
  - LEO Pharma Investigational Site, Frankfurt
  - LEO Pharma Investigational Site, Hamburg
  - LEO Pharma Investigational Site, Langenau
  - LEO Pharma Investigational Site, Lübeck
  - LEO Pharm Investigational Site, Mainz
  - LEO Pharma Investigational Site, Münster
- Greece (3):
  - LEO Pharma Investigational Site, Athens
  - LEO Pharma Investigational Site, Piraeus
  - LEO Pharma Investigational Site, Thessaloniki
- Hungary (2):
  - LEO Pharma Investigational Site, Debrecen
  - LEO Pharma Investigational Site, Orosháza
- Italy (3):
  - LEO Pharma Investigational Site, Brescia
  - LEO Pharma Investigational Site, Napoli
  - LEO Pharma Investigational Site, Padua
- Poland (6):
  - LEO Pharma Investigational Site, Iwonicz-Zdrój
  - LEO Pharma Investigational Site, Lodz
  - LEO Pharma Investigational Site, Poznan
  - LEO Pharma Investigational Site, Skierniewice
  - LEO Pharma Investigational Site, Warsaw
  - LEO Pharma Investigational Site, Wroclaw
- Spain (6):
  - LEO Pharma Investigational Site, Alicante
  - LEO Pharma Investigational Site, Barcelona
  - LEO Pharma Investigational Site, Granada
  - LEO Pharma Investigational Site, Madrid
  - LEO Pharma Investigational Site, Pontevedra
  - LEO Pharma Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across countries in Europe (Belgium, Germany, Hungary, Italy, Poland, Spain) from December 2022 to May 2023 when the study was early terminated.
Pre-assignment Details: In the 12 weeks Induction Period (Week 0 to Week 12) participants were assigned to brodalumab, ustekinumab or placebo. This was followed by a Maintenance Period of 40 weeks (Week 12 to Week 52) where those receiving ustekinumab or brodalumab continued with the same medication whereas participants on placebo were switched to either brodalumab or ustekinumab.
Groups:
- Brodalumab: Participants were randomised to receive brodalumab subcutaneously (SC) at Weeks 0, 1, 2, and then every 2 weeks until week 50. The dose was determined by the participant's body weight. Participants weighing 30 to <70 kg received 140 mg brodalumab, participants weighing ≥70 kg received 210 mg brodalumab. Participants randomised at Week 0 to brodalumab would have continued with the allocated treatment until Week 52.
- Ustekinumab: Participants were randomised to receive ustekinumab SC at Week 0 and 4, and then every 12 weeks until Week 50. The dose was determined by the participant's body weight. Participants weighing 30 to <60 kg received 0.75 mg ustekinumab per kg body weight. Participants weighing ≥60 and ≤100 kg received 45 mg ustekinumab, and those weighing >100 kg received 90 mg ustekinumab. Participants randomised at Week 0 to ustekinumab would have continued with the allocated treatment until Week 52.
- Placebo/Brodalumab: Participants were randomised to receive placebo at Weeks 0, 1, 2, 4, 6, 8, and 10. Following the initial 12 Weeks of placebo, participants received brodalumab at Weeks 12, 13, 14, and every 2 weeks thereafter, with the last brodalumab dose administered at Week 50. The doses were body weight-dependent, participants weighing 30 to <70 kg received 140 mg brodalumab or 1.0 mL placebo. Participants weighing ≥70 kg received 210 mg brodalumab or 1.5 mL placebo.
- Placebo/Ustekinumab: Participants were randomised to receive placebo at Weeks 0, 1, 2, 4, 6, 8, and 10. Following the initial 12 Weeks of placebo, participants received ustekimumab at Weeks 12, 16, 28, and 40. Doses of ustekimumab were body weight-dependent, participants weighing 30 to <60 kg received 0.75 mg/kg. Participants weighing ≥60 and ≤100 kg received 45 mg ustekinumab, and those weighed >100 kg received 90 mg ustekinumab.
Period: Overall Study
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Started | 2 | 6 | 2 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 2 | 6 | 2 | 2
Not completed — Study early termination | 2 | 5 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to low enrollment, baseline data are not reported to protect participant confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index (PASI) 75 Response, Assessed at Week 12.
Description: PASI 75 response is defined as having at least 75% improvement in PASI score from baseline. The severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions, head/neck, trunk, upper extremities, and lower extremities, were assessed according to a severity scale. The extent of psoriasis within each of the 4 body regions was also assessed. This gives a composite score ranging from 0 to 72, with higher values indicating a more severe and/or more extensive condition.
Time Frame: Baseline to Week 12
Population: Participants who completed at Week 12 are included in the overall number of participants analysed. Dataset from the full analysis set (FAS) which includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 1 | 0 | 0 | 1
Participants | NA — Due to early termination, only 2 participants completed Week 12 and therefore, no data is reported to maintain participant confidentiality. |  |  | NA — Due to early termination, only 2 participants completed Week 12 and therefore, no data is reported to maintain participant confidentiality.

2. Secondary Outcome: Static Physician's Global Assessment (sPGA) Score of 0 or 1, Assessed at Week 12.
Description: The sPGA is an instrument used in clinical trials to rate the severity of the participant's global psoriasis and is based on a 6-point scale ranging from 0 (clear) to 5 (very severe). The number of participants achieving a score of 0 (clear) or 1 (almost clear) was assessed.
Time Frame: Week 12
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: sPGA Score of 0, Assessed at Week 12.
Description: as for outcome 2
Time Frame: Week 12
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: PASI 90 Response, Assessed at Week 12.
Description: PASI 90 response is defined as having at least 90% improvement in PASI score from baseline. The severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions, head/neck, trunk, upper extremities, and lower extremities, will be assessed according to a severity scale. The extent of psoriasis within each of the 4 body regions will also be assessed. This gives a composite score ranging from 0 to 72, with higher values indicating a more severe and/or more extensive condition.
Time Frame: Baseline to Week 12
Population: Participants who completed at Week 12 are included in the overall number of participants analysed. Dataset from the FAS which includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 1 | 0 | 0 | 1
Participants | NA — Due to early termination, only 2 participants completed Week 12 and therefore, no data is reported to maintain participant confidentiality. |  |  | NA — Due to early termination, only 2 participants completed Week 12 and therefore, no data is reported to maintain participant confidentiality.

5. Secondary Outcome: PASI 100 Response, Assessed at Week 12.
Description: PASI 100 response is defined as having at least 100% improvement in PASI score from baseline. The severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions, head/neck, trunk, upper extremities, and lower extremities, will be assessed according to a severity scale. The extent of psoriasis within each of the 4 body regions will also be assessed. This gives a composite score ranging from 0 to 72, with higher values indicating a more severe and/or more extensive condition.
Time Frame: Baseline to Week 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 1 | 0 | 0 | 1
Participants | NA — Due to early termination, only 2 participants completed Week 12 and therefore, no data is reported to maintain participant confidentiality. |  |  | NA — Due to early termination, only 2 participants completed Week 12 and therefore, no data is reported to maintain participant confidentiality.

6. Secondary Outcome: Children's Dermatology Life Quality Index (CDLQI) Total Score of 0 or 1, Assessed at Week 12.
Description: CDLQI consists of 10 items addressing the child's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point scale ranging from 0 (not at all) to 3 (very much). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Time Frame: Week 12
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Family Dermatology Life Quality Index (FDLQI) Total Score of 0 or 1, Assessed at Week 12.
Description: FDLQI consists of 10 items addressing the participant's relative perception of the impact of the participant's skin disease on various aspects of his/her quality of life over the last month such as: emotional distress, social life, job and leisure activities, physical well-being, time spent on helping the subject with e.g., treatment procedures, extra housework, and routine household expenditure. Each item is scored on a 4-point scale ranging from 0 (not at all) to 3 (very much). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Time Frame: Week 12
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Overall Number of Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in subjects or clinical investigation participants administered a pharmaceutical product, which does not necessarily have to have a causal relationship with this treatment. A serious AE is defined as any AE that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect or important medical events that do not meet the preceding criteria but based on appropriate medical judgment may jeopardize the patient or may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: Up to approximately 5 months
Population: Dataset from the safety analysis set (SAS) which includes all participants who received at least 1 dose of IMP.
Measure: Number; unit: Adverse events
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 2 | 6 | 2 | 2
Adverse events
  Any AEs | 4 | 5 | 0 | 3
  Any AEs related to IMP | 0 | 3 | 0 | 0

9. Secondary Outcome: Presence of Anti-drug Antibodies, Assessed at Weeks 4, 16, and 52.
Description: Number of participants with a positive post-baseline anti-drug antibody result at weeks 4, 16, and 52.
Time Frame: Week 4, Week 16, and Week 52
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Serum Concentration of Interleukin-17, Assessed at Weeks 8, 12, and 52.
Description: Number of participants with detectable levels of Interleukin-17 at weeks 8, 12, and 52.
Time Frame: Week 8, Week 12, and Week 52
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Blood Levels of T-cell Subsets (CD4+ and CD8+), Assessed at Weeks 8, 12, and 52.
Description: Number of participants with detectable levels of T-cell subsets at weeks 8, 12, and 52.
Time Frame: Week 8, Week 12, and Week 52
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Serum Concentrations of Brodalumab, Assessed at Weeks 4, 8, 10, 12, 16, 22, and 52.
Description: Number of participants with detectable levels of brodalumab at weeks 4, 8, 10, 12, 16, 22, and 52.
Time Frame: Week 4, Week 8, Week 10, Week 12, Week 16, Week 22, and Week 52
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Anti-tetanus Toxoid Antibodies ≥0.1 IU/mL, Assessed at Week 12.
Description: Number of participants with detectable levels of anti-tetanus toxoid antibodies at weeks 12.
Time Frame: Week 12
Population: Due to early termination, data was not collected
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 5 months
Description: Data from the safety analysis set, all participants received at least 1 dose of the investigational medicinal product.
Arm/Group | Brodalumab | Ustekinumab | Placebo/Brodalumab | Placebo/Ustekinumab
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 3/6 | 0/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brodalumab (N=2) | Ustekinumab (N=6) | Placebo/Brodalumab (N=2) | Placebo/Ustekinumab (N=2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression rating scale score increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT04305327/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT04305327/SAP_003.pdf